CLINICAL TRIAL: NCT05961670
Title: Application of Lung Near-Infrared Spectroscopy (NIRS) During Invasive and Non-Invasive Ventilation and Pre- and Post-Surfactant Administration in Preterm Infants
Brief Title: Application of Lung Near-Infrared Spectroscopy (NIRS) in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Keck School of Medicine of USC (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Manoj Biniwale, Associate Professor of Pediatrics, Keck School of Medicine of USC
Other Study IDs: 13184
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Neer Infrared Spectroscopy — Premature infants will be studied with brain and lung NIRS before and after surfactant administration

SUMMARY:
Premature infants are more likely to develop hypoxemia after birth often requiring invasive and Non-Invasive Mechanical ventilation and surfactant therapy to improve alveolar gas exchange and oxygen transport. Near-infrared spectroscopy (NIRS) has been used to detect pulmonary regional oxygen saturation (rpSO 2 ) as well as cerebral regional oxygen saturation (rcSO2 ) and evaluate the oxygenation state of the lung and brain. This is a prospective observational study to evaluate utility of rpSO2 and compare it with rcSO2 in preterm infants born between 23-32 weeks of gestation receiving noninvasive ventilation and surfactant treatment. Enrolled patients will be continuously studied with placement of NIRS monitor using cerebral sensor (INVOS™) for 6 hrs and 15 min before and after surfactant administration. Pulmonary regional oxygen saturation (rpSO2) with a sampling interval of 6 s will be followed for 6hrs.

ELIGIBILITY:
Inclusion Criteria:

Infants born between 23-32 weeks of gestation admitted to the Neonatal Intensive Care Unit with respiratory distress receiving non-invasive ventilation and requiring Surfactant Replacement Therapy.

Exclusion Criteria:

Neonates with no need for respiratory support/Surfactant. Neonates with congenital malformations.

Ages: 1 Hour to 24 Hours | Sex: All
Age Groups: Child
Study Population: Inborn premature infants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
rpSO2 before and after surfactant therapy | 6 hours
  brain and lung rpSO2 will be compared before and after surfactant administration

SECONDARY OUTCOMES:
variations on rpSO2 and rcSO2 during changes in ventilation modes | 6 hours
  Will evaluate for variations with various ventilation modes
correlation between rpSO2L and SpO2/FiO2 ratio, a/APO2, and O.I | 6 hours
  Correlation will be assessed between rpSO2 and other ratios

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles General Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided